CLINICAL TRIAL: NCT02236845
Title: Pilot, Randomized, Cross-over Study to Evaluate Safety and Clinical Effect of Lacrima Medical Device in Patients With Chronic Insomnia
Brief Title: Pilot Study to Clinical Evaluate Lacrima Medical Device in Insomnia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lacrima Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LM002
Record Dates: First submitted 2014-09-06; First posted 2014-09-11 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Insomnia
Keywords: Insomnia, medical device, sleep latency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lacrima medical active device (Experimental)
  Interventions: Device: Lacrima Medical Device and sham comparator
- Lacrima medical sham device (Sham Comparator)
  Interventions: Device: Lacrima Medical Device and sham comparator

INTERVENTIONS:
Device: Lacrima Medical Device and sham comparator

SUMMARY:
The study will assess the safety, tolerability and feasibility of Lacrima investigational medical device vs. sham device in adult patients with chronic Insomnia

ELIGIBILITY:
Main Inclusion Criteria:

1. Adult subjects, 18 years of age and older at screening
2. Diagnosis of primary insomnia based on International Classification of Sleep Disorders, revision no 2
3. Total score of Pittsburgh Sleep Quality questionnaire is > 5
4. Latency to persistent sleep is > 30 minutes based on Pittsburgh questionnaire
5. Able to understand and provide written informed consent

Main Exclusion Criteria:

1. Patients using any pharmacological treatments for insomnia for 14 days
2. Patients currently using stimulants drugs 7 days
3. Patients currently using antidepressants causing sleepiness
4. Patients who are unable to commit to avoid consumption alcohol during the study
5. Patients who are unable to commit to avoid consumption caffeine after 12 pm
6. Patients who have a clinical significant or unstable medical or surgical condition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events | Up to 37 days

SECONDARY OUTCOMES:
Change in sleep latency time based on sleep actigraph | 28 days

OTHER OUTCOMES:
Change in sleep latency time based on sleep diaries | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel